CLINICAL TRIAL: NCT02517151
Title: Effects of Iron Therapy in Patients With Chronic Fatigue and IBD
Brief Title: Iron Supplementation in Inflammatory Bowel Disease (IBD) Patients With Chronic Fatigue
Acronym: MICI_2011-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 868
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Fatigue; Inflammatory Bowel Disease
Keywords: iron; fatigue; crohn's disease; ulcerative colitis; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue; Crohn Disease; Colitis, Ulcerative | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Experimental): 200 mg in normal saline (NS) 100 ml administered i.v. at day 0 and then every 4 weeks up to week 24.
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): normal saline (NS) 100 ml administered i.v. at day 0 and then every 4 weeks up to week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose
  Other Names: Ferinject
  Arms: Ferric carboxymaltose
Drug: Placebo
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
A phase 2, randomized, placebo controlled trial evaluating the effects of n intravenous iron supplementation on chronic fatigue in IBD patients with controlled disease.

DETAILED DESCRIPTION:
The study will evaluate a 6 months therapy with intravenous ferric carboxymaltose.

Patients will undergo a 2-5 days screening period and then will be treated every 4 weeks with iron supplementation/placebo.

At every visit, hematology and blood iron levels will be evaluated. Treatment will be temporarily stopped in case of either Hemoglobin levels above 16 g/dl or ferritin above 800 ng/ml (level decreased to 500 ng/ml in case of Transferrin-Iron Saturation Percentage above 50%).

Study team will be composed of blinded and unblinded personnel and dedicated infusion devices will be used to ensure the double blinding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis or Crohn's Disease established at least 6 months prior to Day 1 by endoscopy and/or imaging
* At least 6 months of clinical remission (Harvey Bradshaw Index ≤5; Mayo clinical score ≤ 2)
* Therapy with mesalamine, immunosuppressors or anti-tumor necrosis factor alpha (TNFα) at stable doses for at least 3 months prior enrollment; steroids are not permitted from 6 months prior baseline
* Chronic fatigue symptoms (MFI-20>13)
* Iron deficiency: ferritin < 100 microg/l or < 300 microg/l in case of Transferrin-Iron Saturation Percentage (TSAT) <20%
* Women of childbearing potential must have a negative serum pregnancy test before enrollment.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Known hypersensibility to active principle or excipients
* Pregnant or lactating women
* Clinically active IBD (Harvey Bradshaw Index >6; Mayo clinical score >3 or C-Reactive Protein >2.5 mg/L
* Renal failure (eGFR<60)
* History of adrenal insufficiency
* History of autoimmune diseases
* History of malignancies
* Depression
* Any current or recent signs or symptoms of viral infectious diseases
* Recent psycho-traumatic events
* Hemoglobin levels < 12.5 g/dl (men) or <11.5 g/dL (women)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
chronic fatigue remission | Week 24
  Multidimensional fatigue inventory (MFI-20) <13

SECONDARY OUTCOMES:
Chronic fatigue reduction | Week 24
  MFI-20 reduction of at least 4 points (absolute MFI-20>13)
chronic fatigue remission | Week 12
  MFI-20 <13
Anxiety evaluation | week 4, week 12, week 24
  State-Trait Anxiety Inventory (STAI)Y1 and STAI Y2 values
Depression evaluation | week 4, week 12, week 24
  BECK DEPRESSION INVENTORY (BDI-II) values
Quality of life | week 4, week 12, week 24
  Inflammatory Bowel Disease Questionnaire (IBDQ) values

CONTACTS AND LOCATIONS:
Locations (1):
- IBD Center, Rozzano, MI, Italy